CLINICAL TRIAL: NCT05342766
Title: Nutritia de Precizie
Brief Title: Precision Nutrition
Acronym: NP
Status: Completed | Type: Observational
Sponsor: Shape Divine Center SRL (Other)
Collaborators: SmartepigenetX SRL (Unknown); Advanced Nutrigenomics LLC (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2022-0101-21493351
Record Dates: First submitted 2022-04-17; First posted 2022-04-25 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2022-04

CONDITIONS: Nutrient Deficiency
Keywords: Genotypes; Nutrient intakes; Nutrient plasma levels

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1: Half of participants (healthy M and F, no children), randomly assigned. Group assignment will balance sex distribution. Nutrigenetic testing will be performed prior to intervention. Participants will work with a registered dietician, who will assess their current nutrient intakes and corresponding nutrient plasma values (T0). Target nutrient intakes will be determined based on nutrigenetic assessment. Participants undergo a nutrition intervention (first 3 months, Intervention 1), in which the difference between actual intakes and nutrigenetically-recommended intakes will be provided using supplements. At the end of Intervention 1 (T1), nutrient plasma values will be measured. After a wash-out period (3 months, no supplementation), nutrient plasma levels will be measured (T2), and a second intervention (3 months, Intervention 2) will consist of supplements administered according to EFSA recommended levels. At the end of Intervention 2, plasma nutrient levels will be measured (T3).
  Interventions: Dietary Supplement: Nutrigenetic
- Group 2: Half of participants (healthy M and F, no children), randomly assigned. Group assignment will balance sex distribution. Nutrigenetic testing will be performed prior to intervention. Participants will work with a registered dietician, who will assess their current nutrient intakes and corresponding nutrient plasma values (T0). Target nutrient intakes will be determined based on nutrigenetic assessment. Participants undergo a nutrition intervention (first 3 months, Intervention 1), in which the difference between actual intakes and EFSA-recommended intakes will be provided using supplements. At the end of Intervention 1 (T1), nutrient plasma values are measured. After a wash-out period (3 months, no supplementation), nutrient plasma levels will be measured (T2), and a second intervention (3 months, Intervention 2) will consist of supplements administered according to targets recommended by nutrigenetic testing. At the end of Intervention 2, plasma nutrient levels will be measured (T3).
  Interventions: Dietary Supplement: Nutrigenetic

INTERVENTIONS:
Dietary Supplement: Nutrigenetic — Each grup will receive two interventions ("Nutrigenetic" and "Standard"), in a cross-over design (3 months each), spaced by a wash-out period (3 months).
  Other Names: Standard

SUMMARY:
Determine the relationship between relevant genotypes and nutrient plasma levels, with the aim to normalize such levels using a nutritional intervention.

(Original text in Romanian language: Caracterizarea precisa a relatiei dintre variatiile genetice si nivelul de nutrienti din sange/plasma/ser, in scopul de a defini modul in care aportul alimentar poate normaliza aceste nivele.)

DETAILED DESCRIPTION:
1. Define plasma levels prediction formulas for each involved nutrient, based on relevant genotypes;
2. Characterize the roles that food intakes may have in the alteriations of such plasma levels, depending on genotype structure;
3. Based on clinical data, create predictive equations using dependent variables (genotypes) in order to define optima nutrient intakes;
4. (Secondary aim): compare the efficacy of a nutrigenetic-based intervention with a non-nutrigenetic intervention (classical approach).

(Original text in Romanian language:

1. Definirea unor formule de predictie a nivelelor din sange, in functie de variatiile genetice;
2. Caracterizarea rolului pe care aportul alimentar de nutrienti il are in modularea acestor valori, in contextul variatiilor genetice.
3. Gasirea unor formule de predictie in care variabilele independente (variatii genetice si combinatii ale acestora) sa defineasca necesarul de nutrienti pentru a normaliza valorile sangvine ale acestor nutrienti.
4. (Obiectiv secundar): compararea eficacitatii unei interventii nutrigenetice fata de o interventie clasica nutritionala (non-nutrigenetica).)

ELIGIBILITY:
Inclusion Criteria:

* healthy adults

Exclusion Criteria:

* any pathology

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy adults
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
blood/serum nutrient levels | 3 months
  nutrients as follows:
  * ALA
  * LA
  * A
  * D
  * E
  * K
  * Riboflavina
  * Niacina
  * Folati
  * B12
  * Calciu
  * Magneziu
  * Seleniu
  * Zinc
  Each nutrient (having different system of measure) will be considered as a separate outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Shape Divine SRL, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: No
Publication of the results